CLINICAL TRIAL: NCT04261361
Title: A Randomized Controlled Trial of Community-based Cognitive Behavioral Therapy for Type 2 Diabetes in Hong Kong
Brief Title: Community-based Cognitive Behavioral Therapy for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Au May-lan Alma, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HMRFCBCBT
Record Dates: First submitted 2017-05-22; First posted 2020-02-07 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Depression
Keywords: telephone follow-up; sustainability; cognitive behavioural therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBCBT intervention (Experimental): 1. Adherence counseling
  2. Psycho-education package
  3. The intervention program consists of three components: 1) eight weekly sessions of face-to-face interventions, 2) four weekly consolidation individual telephone calls and 3) three monthly individual follow-up phone calls.
  Interventions: Behavioral: CBCBT intervention; Behavioral: Adherence counseling; Behavioral: Psycho-education package
- enhanced treatment as usual (ETAU) (Active Comparator): 1. Adherence counseling;
  2. Psycho-education package;
  3. To maintain some control over the contact time, we will give them 4 bi-weekly individual phone calls of about 10 minutes each while the CBCBT intervention group is having their 8 weeks of face-to-face group sessions.
  Interventions: Behavioral: Adherence counseling; Behavioral: Psycho-education package

INTERVENTIONS:
Behavioral: CBCBT intervention — 8 group CBT sessions and 4 weekly follow-up calls
  Other Names: CBT
  Arms: CBCBT intervention
Behavioral: Adherence counseling — All participants in both CBCBT and ETAU groups will have one session of Life-Steps, a stand-alone CBCBT intervention designed to improve adherence to medical recommendations and individualized DM self-management goals.
Behavioral: Psycho-education package — Printed materials of a DM self-management education program will be delivered to both the CBCBT and ETAU groups.

SUMMARY:
Objectives: The aim of the study is evaluate the efficacy of a telephone assisted cognitive behavioral therapy for adherence (CBCBT) in type 2 diabetes.

Hypothesis: CBCBT will primarily reduce depressive symptoms and improve glycemic control and secondarily, improve adherence and self-care and reduce diabetes-specific distress.

Design and subjects: This is a prospective randomized two-armed intervention study. One hundred sixty eight participants will be recruited from five sites covering the following clusters: New Territories East, Kowloon East and Hong Kong West.

Intervention: The CBT protocol (Safren et al., 2013) will be used in the intervention. Specific components include: 1) introducing CBT for behavior change, 2) increasing pleasurable activities and mood monitoring, 3) cognitive restructuring, 4) problem-solving in self-care and 5) relaxation training. To maximize accessibility, eight sessions will be delivered face-to-face in group setting and the other four sessions will be delivered by telephone. Three monthly follow-up telephone calls will be made to consolidate treatment gains.

Main outcome measures: Primary outcomes include the Beck Depression Inventory and glycemic control. Secondary outcomes include self-care and diabetes-specific distress.

Data analysis: Treatment outcomes will be assessed by Repeated Measures ANOVA and also Intention to Treat Analysis. Regression models will be used to estimate effect sizes and associations among variables.

Expected results: CBCBT would significantly reduce depressive symptoms and improve glycemic control. With secondary outcomes, CBCBT will improve self-care and reduce diabetes-specific distress.

DETAILED DESCRIPTION:
A community-based CBCBT is tested for patients living with diabetes(DM) and subclinical depression. The program includes both face-to-face group sessions and individual telephone sessions. The aim of the current study is to evaluate the efficacy of a mixed mode CBCBT in reducing depressive symptoms and enhancing adherence among adults with DM and subclinical depression. The intervention program consists of three components: 1) eight weekly sessions of face-to-face interventions, 2) four weekly consolidation individual telephone calls and 3) three monthly individual follow-up phone calls.

This is a prospective randomized two-armed intervention study. The CBCBT intervention will be compared with enhanced treatments usual (ETAU) using a single blinded randomized design. The intervention will be delivered by qualified health care professional (e.g. clinical psychology/ social worker/ nurse counsellor) who have had some training in CBCBT in the initial training.

ELIGIBILITY:
Inclusion Criteria:

* Patients have to meet the following criteria: 1) aged between 25 to 60 years; 2) living with Type 2 DM, 3) community dwelling, 4) independent in their activities of daily living as indicated on the Barthel Index and 5) obtained on screening a score of 5 to 9 on the Patient Health Questionnaire Depression Scale (PHQ-9).

Exclusion Criteria:

* Patients will be excluded by a clinician/ investigator for major depression within the past 6 months, lifetime history of other psychiatric disorder including psychosis, schizophrenia ad bipolar affective disorder, serious suicidal risk, alcohol or substance abuse and medical illnesses with prognosis of less than 12 months to live (as identified by reviewing their medical history), already taking medication or receiving psychological intervention for depressive disorders or related symptom, bedridden, having memory loss, not being able to understand or communicate in Chinese language, or refusing to give consent.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Change from baseline through study completion, an average of 24 weeks
  The Beck Depression Inventory (BDI-I) assesses cognitive, behavioral and somatic symptoms of depression.
Glycemic control | Change from baseline through study completion, an average of 24 weeks
  Glycated haemoglobin (HbA1c) is used to measure glycemic control

SECONDARY OUTCOMES:
The Summary of DM Self-care Activities Questionnaire (SDSCA) | Change from baseline through study completion, an average of 24 weeks
  The revised 11-item SDSCA assess aspects of diabetes self-management that includes diet, exercise, self-monitoring of blood-glucose, foot care, and smoking in the past 7 days (0-7 points) by self-reported frequency.
DM-specific distress | Change from baseline through study completion, an average of 24 weeks
  The DM Distress Scale (DDS) is a 17-item self-administered questionnaire identifying four domains of DM-related distress: emotional burden, physician-related distress, regimen related distress, and interpersonal distress

CONTACTS AND LOCATIONS:
Overall Officials: Alma Au, PhD, Principal Investigator — Applied Social Sciences, Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Applied Social Sciences, Hong Kong Polytechnic University, Hong Kong
  - Institute of Active Ageing, Kowloon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldney RD, Phillips PJ, Fisher LJ, Wilson DH. Diabetes, depression, and quality of life: a population study. Diabetes Care. 2004 May;27(5):1066-70. doi: 10.2337/diacare.27.5.1066. PMID 15111522
- [Background] Ali S, Stone MA, Peters JL, Davies MJ, Khunti K. The prevalence of co-morbid depression in adults with Type 2 diabetes: a systematic review and meta-analysis. Diabet Med. 2006 Nov;23(11):1165-73. doi: 10.1111/j.1464-5491.2006.01943.x. PMID 17054590
- [Background] Gonzalez JS, Shreck E, Psaros C, Safren SA. Distress and type 2 diabetes-treatment adherence: A mediating role for perceived control. Health Psychol. 2015 May;34(5):505-13. doi: 10.1037/hea0000131. Epub 2014 Aug 11. PMID 25110840
- [Background] Cully JA, Breland JY, Robertson S, Utech AE, Hundt N, Kunik ME, Petersen NJ, Masozera N, Rao R, Naik AD. Behavioral health coaching for rural veterans with diabetes and depression: a patient randomized effectiveness implementation trial. BMC Health Serv Res. 2014 Apr 28;14:191. doi: 10.1186/1472-6963-14-191. PMID 24774351
- [Background] Glasgow RE, Nelson CC, Strycker LA, King DK. Using RE-AIM metrics to evaluate diabetes self-management support interventions. Am J Prev Med. 2006 Jan;30(1):67-73. doi: 10.1016/j.amepre.2005.08.037. PMID 16414426
- [Background] Nan H, Au A, Sum R, et al. Effect of family support intervention in diabetic retinopathy with depressive symptoms: a randomized clinical trial in Hong Kong. The 10th International Diabetes Federation-Western Pacific Congress. Suntec Singapore: International Diabetes Federation-Western Pacific Congress, 2014:ABS-1807.
- [Background] Zhang Y, Ting R, Lam M, Lam J, Nan H, Yeung R, Yang W, Ji L, Weng J, Wing YK, Sartorius N, Chan JCN. Measuring depressive symptoms using the Patient Health Questionnaire-9 in Hong Kong Chinese subjects with type 2 diabetes. J Affect Disord. 2013 Nov;151(2):660-666. doi: 10.1016/j.jad.2013.07.014. Epub 2013 Jul 31. PMID 23938133
- [Background] Au A, Gallagher-Thompson D, Wong MK, Leung J, Chan WC, Chan CC, Lu HJ, Lai MK, Chan K. Behavioral activation for dementia caregivers: scheduling pleasant events and enhancing communications. Clin Interv Aging. 2015 Mar 26;10:611-9. doi: 10.2147/CIA.S72348. eCollection 2015. PMID 25848237
- [Background] Katon W, Unutzer J, Fan MY, Williams JW Jr, Schoenbaum M, Lin EH, Hunkeler EM. Cost-effectiveness and net benefit of enhanced treatment of depression for older adults with diabetes and depression. Diabetes Care. 2006 Feb;29(2):265-70. doi: 10.2337/diacare.29.02.06.dc05-1572. PMID 16443871
- [Background] Chan BS, Tsang MW, Lee VW, Lee KK. Cost of Type 2 Diabetes mellitus in Hong Kong Chinese. Int J Clin Pharmacol Ther. 2007 Aug;45(8):455-68. doi: 10.5414/cpp45455. PMID 17725179
- [Background] Hermanns N, Caputo S, Dzida G, Khunti K, Meneghini LF, Snoek F. Screening, evaluation and management of depression in people with diabetes in primary care. Prim Care Diabetes. 2013 Apr;7(1):1-10. doi: 10.1016/j.pcd.2012.11.002. Epub 2012 Dec 30. PMID 23280258
- [Result] Safren SA, Gonzalez JS, Wexler DJ, Psaros C, Delahanty LM, Blashill AJ, Margolina AI, Cagliero E. A randomized controlled trial of cognitive behavioral therapy for adherence and depression (CBT-AD) in patients with uncontrolled type 2 diabetes. Diabetes Care. 2014;37(3):625-33. doi: 10.2337/dc13-0816. Epub 2013 Oct 29. PMID 24170758